CLINICAL TRIAL: NCT01737983
Title: Lactobacillus Reuteri Reduces Pulmonary Exacerbations and Upper Respiratory Tract Infections in CF Patients With Mild-to-moderate Lung Disease. LR Administration Might Have a Beneficial Effect on the Disease Course of Cystic Fibrosis.
Brief Title: Effect of Lactobacillus Reuteri in Cystic Fibrosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda Policlinico Umberto I (Other)
Responsible Party: Principal Investigator, Giovanni Di Nardo, MD, Azienda Policlinico Umberto I
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: lactobacillus reuteri in fc
Record Dates: First submitted 2012-07-12; First posted 2012-11-30 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: CYSTIC FIBROSIS
Keywords: cystic fibrosis; probiotics; Lactobacillus reuteri
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactobacillus reuteri (LR) ATCC55730 (Experimental): The tested probiotic, Lactobacillus reuteri, was administered in 5 drops per day (10^10 colony-forming units) for 6 months
  Interventions: Dietary Supplement: Lactobacillus reuteri
- placebo (Placebo Comparator): The placebo was packed in identical bottles, had the same color, weight, smell, and taste of the probiotic formulation for 6 months During the test period, patients were not allowed to consume any other product that contained probiotics or prebiotics
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri — Lactobacillus reuteri was administered in 5 drops per day (10^10 colony-forming units) for 6 months.
  Other Names: (LR) ATCC55730
  Arms: Lactobacillus reuteri (LR) ATCC55730
Dietary Supplement: placebo — The placebo was packed in identical bottles, had the same color, weight, smell, and taste of the probiotic formulation, was administered in 5 drops per day
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate in patients with cystic fibrosis the effect of Lactobacillus Reuteri (LR) on the rate of respiratory exacerbations and of the infections of both upper respiratory and gastrointestinal tracts.

DETAILED DESCRIPTION:
The hallmarks of cystic fibrosis (CF) are recurrent severe and destructive pulmonary inflammation and infection, beginning in early childhood and leading to morbidity and mortality due to respiratory failure. During the disease, most children become colonized with Pseudomonas aeruginosa (PA) and undergo progressive impairment of respiratory function. Therefore, patients colonized with Pseudomonas are at increased risk for pulmonary infections and persistent inflammation and have a decrease in survival rate. In an attempt to reduce the rate and severity of pulmonary exacerbations, children with CF are put on heavy load of antibiotics.

Intestinal inflammation is another typical finding in CF patients and gut bacterial overgrowth may be present.

Probiotics are live bacteria administered orally, successfully used in children with acute gastroenteritis, as well as in preventing and treating atopic diseases in children. In addition, probiotics have been used as adjuvant therapy in patients with pouchitis and inflammatory bowel diseases. Interestingly, probiotic supplementation is able to reduce the incidence of fever, child care absences, antibiotic prescription and to prevent nosocomial gastrointestinal and respiratory infections. The effect of probiotics may be through improvement of intestinal barrier function and modulation of immune response. The latter mechanism could well explain the clinical effects of probiotics observed in extraintestinal diseases.

ELIGIBILITY:
Inclusion Criteria:

* Forced expiratory volume in the 1st second (FEV1) > 70%.
* No inhaled or systemic steroids.
* No anti-inflammatory drugs, antileukotrienes and mast cell membrane stabilizers.
* No serious organ involvement.

Exclusion Criteria:

* History of pulmonary exacerbation or upper respiratory infection in the previous two months.
* Changes in medications in the past two months.
* History of hemoptysis in the past two months.

Ages: 6 Years to 42 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 61 (Actual)
Dates: Start 2009-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Efficacy | 6 months of observation
  Evaluate number of episodes of pulmonary exacerbations that were diagnosed by increase in pulmonary symptoms and airway secretions requiring oral or intravenous antibiotics.
Efficacy | 6 months of observation
  Evaluate number of hospital admissions required for pulmonary exacerbations in the two groups.
efficacy | 6 months of observation
  Evaluate number of gastrointestinal and upper respiratory tract infections.
efficacy | 6 months of observation
  Evaluate duration of hospital admissions required for pulmonary exacerbations in the two groups.

SECONDARY OUTCOMES:
efficacy | 6 months of observation
  Evaluate change in qualitative sputum bacteria;
efficacy | 6 months of observation
  Evaluate change in fecal calprotectin concentration.
efficacy | 6 months of observation
  Evaluate interleukin 8 levels in plasma and induced sputum.
efficacy | 6 months of observation
  Evaluate change in quantitative sputum bacteria;
efficacy | 6 months of observation
  Evaluate tumor necrosis factor α levels in plasma and induced sputum.

CONTACTS AND LOCATIONS:
Locations (1):
- Dipartimento di pediatria e neuropsichiatria Policlinico Umberto l "Università di Roma la Sapienza", Roma, Italy

REFERENCES:
- [Derived] Di Nardo G, Oliva S, Menichella A, Pistelli R, De Biase RV, Patriarchi F, Cucchiara S, Stronati L. Lactobacillus reuteri ATCC55730 in cystic fibrosis. J Pediatr Gastroenterol Nutr. 2014 Jan;58(1):81-6. doi: 10.1097/MPG.0000000000000187. PMID 24121143